CLINICAL TRIAL: NCT05664178
Title: Remote Resistance Exercise Powering Survivors - Gastrointestinal Oncology (Remote REPS - GI)
Brief Title: Remote Resistance Exercise Powering Survivors - Gastrointestinal Oncology
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-21742; 1K22CA262352-01 (NIH)
Record Dates: First submitted 2022-12-09; First posted 2022-12-23 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Cancer
Keywords: Gastrointestinal Cancer; Remote Resistance Exercise; GI Cancer Stage III; GI Cancer Stage IV; Tele-Resistance Training
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Resistance Training (RT) (Experimental): Participants will be encouraged to perform approximately 30 minutes of resistance training exercises approximately twice per week for 12 weeks. Participants will also be encouraged to perform moderate aerobic exercise at least 3 times per week. Participants will wear a FitBit fitness watch to monitor aerobic exercise.
  Interventions: Behavioral: Tele-Resistance Training
- Usual Care (UC) (No Intervention): Participants randomized to the Usual Care (UC) arm will be provided with information materials outlining resistance training using body weight or basic equipment. Participants will wear a FitBit fitness watch to monitor aerobic exercise.

INTERVENTIONS:
Behavioral: Tele-Resistance Training — Tele-Resistance training sessions will be supervised and guided by a certified exercise trainer via smartphone, tablet or laptop. Exercises will be performed using resistance tubes (Bodylastics Resistance Bands Set) and a connectable bar (Bionic Body Workout Bar) that mimics a weighted barbell when tubes are attached. The tubes provide up to 142 pounds of resistance (adjustable in increments between 3-10 pounds) when simultaneously connected to handles or bar, and multiple tubes can be attached simultaneously. Participants will engage in brief warm up exercises lasting 2-3 minutes prior to each RT session and will rest at least 1 minute between sets of the same exercise to aid muscle recovery. Participants will perform at least 2 sets of 12 repetitions for each of 6 exercises. Including warm up, training sets, and rest, sessions will last approximately 30 minutes. RT will include six target exercises focusing on major muscle groups of the upper body, lower body, and core.
  Arms: Tele-Resistance Training (RT)

SUMMARY:
The purpose of the study is to evaluate a tele-resistance training exercise program for individuals undergoing chemotherapy for advanced upper gastrointestinal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Biopsy-proven upper GI cancer, stage III-IV
* ECOG performance status 0-1
* Treatment plan of chemotherapy with planned return to Moffitt Cancer Center for restaging
* Able to read and speak English fluently
* Capable of providing informed consent

Exclusion Criteria:

* Regular engagement in RT (2x/week targeting all major muscle groups)
* Screen failure for exercise safety based on Physical Activity Readiness Questionnaire (PAR-Q) and Patient-Reported Measurement Information System (PROMIS) screening questions
* Underlying unstable cardiac or pulmonary disease or symptomatic cardiac disease (New York Heart Association functional class III or IV).
* Recent fracture or acute musculoskeletal injury that precludes ability to participate in RT
* Numeric pain rating scale of ≥ 7 out of 10
* Myopathic or rheumatologic disease that impacts physical function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2026-08-22 (Estimated); Study Completion 2026-08-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants that Enroll and Consent - Enrollment Feasibility | Up to 36 Months
  Enrollment will be considered feasible if ≥ 70% of eligible and approached patients actually consent and enroll
Percentage of Participants that Complete Study Assessments - Retention Feasibility | Up to 3 Months
  Retention will be considered feasible if ≥ 70% of participants who complete baseline measures also complete followup measures
Exercise Adherence - Feasibility | Up to 6 Months
  Exercise adherence will be assessed based on performance of prescribed exercise volume, with tele-RT volumes considered feasible if participants perform ≥ 70% of the volume prescribed.
Participant Evaluation of Feasibility and Acceptability - Acceptability | Up to 6 Months
  Participants evaluation of feasibility and acceptability will be assessed with a questionnaire, adapted to fit the intervention. The questionnaire includes both Likert Scale and open-ended questions. An item-by-item basis and as average item score, with scores ≥4 ("agree" to "strongly agree") indicating acceptability. Open-ended responses will be analyzed qualitatively to inform intervention improvement.
Participant Self-Reported Musculoskeletal Injuries - Safety | Up to 6 Months
  Participants will be asked to report the following information: type (joint or soft tissue or other), location (specific body part), and cause (description of activity during which injury was incurred). Participants will then rate the injury on a scale of 1-4 (1=not related, 2=unlikely related, 3=likely related, 4=definitely related). The severity of the injury will be rated on a scale of 1-4 (1=mild/no change in daily activity, 2=some limitation of daily activity, 3=major limitation of daily activity, 4=life threatening). The duration for which daily activities were impacted will be rated on a scale from 1-5 (1=no change, 2=1-3 days, 3=4-7 days, 4=1-2 weeks, 5=more than 2 weeks). The numerator of the variable used to determine program safety will be the number of musculoskeletal injuries that were rated at least a 3 for relatedness to RT (likely related or definitely related) and caused at least some limitation of daily activity lasting more than 3 days.
Participant Muscular Strength - Baseline | At Baseline
  Muscular strength will be measured using four separate 1-repetition maximum (1RM) lifts: chest press, seated row, leg press, and leg extension performed on resistance training machines. If a particular 1RM lift is contraindicated for a given participant (e.g., limited range of motion for a given joint or osteoporosis), the lift will be skipped, or 5-repetition maximum (5RM) will be measured instead of 1RM, and 1RM will be estimated from 5RM.
Participant Muscular Strength - Follow-up | Up to 6 Months
  Muscular strength will be measured using four separate 1-repetition maximum (1RM) lifts: chest press, seated row, leg press, and leg extension performed on resistance training machines. If a particular 1RM lift is contraindicated for a given participant (e.g., limited range of motion for a given joint or osteoporosis), the lift will be skipped, or 5-repetition maximum (5RM) will be measured instead of 1RM, and 1RM will be estimated from 5RM.
Participant Muscular Endurance - Baseline | At Baseline
  Muscular endurance will be measured by the maximum number of repetitions a participant can perform at 70% of the baseline 1-repetition maximum (1RM) for the same four lifts
Participant Muscular Endurance - Follow-up | Up to 6 Months
  Muscular endurance will be measured by the maximum number of repetitions a participant can perform at 70% of the baseline 1-repetition maximum (1RM) for the same four lifts
Participant Skeletal Muscle Index (SMI) - Baseline | At Baseline
  Participants SMI will be measured using Tomovision SliceOMatic software and clinical, computerized tomography (CT) scans from baseline to follow up.
Participant Skeletal Muscle Index (SMI) - Follow-up | Up to 6 Months
  Participants SMI will be measured using Tomovision SliceOMatic software and clinical, computerized tomography (CT) scans from baseline to follow up.
Participant Skeletal Muscle Density (SMD) - Baseline | At Baseline
  Participants SMD will be measured using Tomovision SliceOMatic software and clinical, computerized tomography (CT) scans from baseline to follow up.
Participant Skeletal Muscle Density (SMD) - Follow-up | Up to 6 Months
  Participants SMD will be measured using Tomovision SliceOMatic software and clinical, computerized tomography (CT) scans from baseline to follow up.
Participants Health-Related Quality of Life | Up to 6 Months
  Health-related quality of life will be measured using the Functional Assessment of Cancer Therapy-General (FACT-G)
Participant Fatigue | Up to 6 Months
  Participant fatigue will be measured using the FACT-Fatigue questionnaire (FACT-F)
Participant Physical Functioning | Up to 6 Months
  Participants physical functioning will be measured using the Patient Reported Outcomes Measurement Information System (PROMIS) Physical Functioning Short Form
Participant Chemotherapy-induced peripheral neuropathy (CIPN) | Up to 6 Months
  Participant CIPN will be measured using the European Organization of Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-CIPN twenty-item scale (QLQ-CIPN20)
Participant Self Reported Exercise - Baseline | At Baseline
  Participant self-reported exercise will be measured using a modified Godin Leisure Time Exercise Questionnaire to assess both aerobic and resistance exercise
Participant Self Reported Exercise - Follow-up | Up to 6 Months
  Participant self-reported exercise will be measured using a modified Godin Leisure Time Exercise Questionnaire to assess both aerobic and resistance exercise
Participant Clinicodemographic Characteristics - Baseline | At Baseline
  Participant clinicodemographic characteristics including tumor type and cancer stage, chemotherapy type, sex, age, body mass index, race/ethnicity, and marital status will be collected from participants' electronic medical records.
Participant Clinicodemographic Characteristics - Follow-up | Up to 6 Months
  Participant clinicodemographic characteristics including tumor type and cancer stage, chemotherapy type, sex, age, body mass index, race/ethnicity, and marital status will be collected from participants' electronic medical records.
Participant Treatment Outcome | Up to 6 Months
  Participant relevant treatment outcomes including chemotherapy dose reductions and changes in chemotherapy will be collected from participants' electronic medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Parker, PhD, MPH, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Search — https://moffitt.org/clinicaltrialssearch?DiseaseSite=&q=21742